CLINICAL TRIAL: NCT05056662
Title: Post-Revascularization Optimization and PHysiological Evaluation of intermediaTe Lesions: an FFR-based Single Center Registry
Brief Title: Post-Revascularization Optimization and PHysiological Evaluation of intermediaTe Lesions
Acronym: PROPHET-FFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Maria Leone, MD, Principal Investigator, Head of Chronic Coronary Syndromes Department at Fondazione Policlinico A. Gemelli, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3237
Record Dates: First submitted 2021-07-22; First posted 2021-09-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Ischemic Heart Disease; Angina, Stable; Non ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction; Unstable Angina; Coronary Disease
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Angina, Unstable; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with negative invasive functional evaluation
  Interventions: Diagnostic Test: Invasive functional evaluation with either Pd/Pa, FFR, iFR or contrast FFR
- Group 2: Patients with positive invasive functional evaluation undergoing PCI
  Interventions: Diagnostic Test: Invasive functional evaluation with either Pd/Pa, FFR, iFR or contrast FFR
- Group 3: Patients with positive invasive functional evaluation undergoing PCI and subsequent retest of functional indexes
  Interventions: Diagnostic Test: Invasive functional evaluation with either Pd/Pa, FFR, iFR or contrast FFR

INTERVENTIONS:
Diagnostic Test: Invasive functional evaluation with either Pd/Pa, FFR, iFR or contrast FFR — Enrolled patients will undergo invasive functional evaluation of coronary stenosis followed by percutaneous revascularization if appropriate. Patients in Group 3 will have target lesion re-assessed using either PdPa, FFR, iFR or contrast FFR.

SUMMARY:
PROPHET-FFR is a single center ambispective registry aiming to explore the impact of post-revascularization functional assessment on later outcomes.

DETAILED DESCRIPTION:
PROPHET-FFR is a ambispective observational study enrolling patients that need invasive functional evaluation in the diagnostic workup of coronary artery disease.

Clinical outcomes of patients that undergo functional assessment after PCI will be compared both to patients undergoing PCI without further evaluations and both to patients that will be deferred due to to negative functional evaluation.

Since the observational nature of the study the decision to perform post-PCI physiological assessment will be left to operator's discretion.

In case of post-PCI functional evaluation results that will be deemed as unsatisfactory by the operator further actions can be taken in order to optimize procedural result. The decision on this opportunity as well as the choice of the strategy to adopt are left to operator's discretion.

The primary endpoint of the study is the rate of MACE defined as the composite of spontaneous MI, target vessel failure, cardiac deaths at 24 months. Follow up will be performed by telephone contact and medical records screening at 12, 24 and 36 months.

Moreover data about in-hospital events will be collected including the release of myocardial damage markers, change in Creatinine, and lenght of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* requiring coronary angiography to assess coronary artery disease;
* having at least one angiographically intermediate coronary stenosis (eg. 40%-80%) on any vessel requiring invasive functional assessment using FFR (and/or any other surrogate index)
* being able and legally entitled to give informed consent

Exclusion Criteria:

* history of severe poorly uncontrolled pulmonary disease
* hemodynamic instability during the diagnostic or therapeutic procedures;
* known adenosine intolerance
* need of mechanical circulatory or ventilatory support;
* stage IV chronic kidney disease.
* life expectancy <1 year
* patients gaining indication to surgical revascularization;
* major procedural complications during percutaneous revascularization (cardiac arrest needing cardiopulmonary resuscitation, major bleeding , large iatrogenic coronary dissection, coronary embolization in a main vessel, suspected stroke) making post-PCI functional evaluation unsafe or impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring invasive functional evaluation of epicardial stenosis to guide revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of composite of Major Adverse Cardiovascular Events (MACE) [ Cardiac Death/Myocardial Infarction/Target Vessel Failure (TVF)] | 2 years

SECONDARY OUTCOMES:
Rate of any component of MACE (Cardiac Death/Myocardial Infarction/Target Vessel Failure (TVF)] | 1 year, 3 years, 5 years
Rate of all-cause Death | 1 year, 3 years, 5 years
Rate of recurrent or persistent angina | 1 year, 3 years, 5 years
Percentage of change in angina intensity assessed by shortened Seattle Angina Questionnaire-7 | 1 year, 3 years, 5 years
  A score ranging from 0 to 100, with the higher values associated with less severe symptoms
Rate of cardiac hospitalizations | 1 year, 3 years, 5 years
  Any hospitalization for cardiac causes
absolute and relative change in functional indexes measured before and after any step of the study procedure | intraprocedural
post-procedural troponin level | 24 hours and 48 hours
  ng/L
post-procedural creatinine level | 24 hours and 48 hours
  mg/dL
procedural cost | intraprocedural
  Euro
fluoroscopy time | intraprocedural
  minutes
contrast dose | intraprocedural
  mL
number of stents implanted and balloon used for optimization | intraprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Agostino Gemelli, Rome, RM, Italy

REFERENCES:
- [Derived] Galante D, Migliaro S, Di Giusto F, Anastasia G, Petrolati E, Vicere A, Zimbardo G, Cialdella P, Romagnoli E, Aurigemma C, Burzotta F, Trani C, Martin-Reyes R, Baptista SB, Faria D, Amabile N, Raposo L, Crea F, Leone AM. Age and Vasodilator Response to Different Hyperemic Agents: Adenosine versus Contrast Medium. Rev Cardiovasc Med. 2024 Jul 2;25(7):239. doi: 10.31083/j.rcm2507239. eCollection 2024 Jul. PMID 39139436